CLINICAL TRIAL: NCT01766921
Title: A Phase II, Randomized, Observer-Blind, Multi-Center, Study to Evaluate Safety, Tolerability and Immunogenicity of an Adjuvanted Cell Culture-Derived H5N1 Subunit Influenza Virus Vaccine at Two Different Formulations in Healthy Elderly Subjects.
Brief Title: Safety and Immunogenicity of Two Doses of H5N1 Influenza Vaccine in Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V89_13
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Pandemic H5N1 Influenza
Keywords: Influenza, Pandemic, H5N1, Elderly adults
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- aH5N1c - High dose (Experimental)
  Interventions: Biological: Adjuvanted H5N1 pandemic influenza vaccine
- aH5N1c - Low dose (Experimental)
  Interventions: Biological: Adjuvanted H5N1 pandemic influenza vaccine

INTERVENTIONS:
Biological: Adjuvanted H5N1 pandemic influenza vaccine — Comparison of two doses of aH5N1c vaccine

SUMMARY:
Evaluate Safety, Tolerability and Immune response of adjuvanted H5N1 cell culture derived influenza vaccine in elderly subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy elderly subjects ≥65 years,
2. Individuals willing to provide written informed consent,
3. Individuals in good health,
4. Individuals willing to allow for their serum samples to be stored beyond the study period.

Exclusion Criteria:

1. Individuals not able to understand and follow study procedures,
2. History of any significant illness,
3. History of any serious chronic medical condition or progressive disease,
4. Presence of medically significant cancer,
5. Known or suspected impairment/alteration of immune function,
6. Presence of any progressive or severe neurologic disorder,
7. Presence of any bleeding disorders or conditions that prolongs bleeding time,
8. History of allergy to vaccine components,
9. Receipt of any other investigational product within 30 days prior to entry into the study,
10. History of previous H5N1 vaccination,
11. Receipt of any other type of seasonal vaccination within 2 months prior to entry into the study,
12. Receipt of any other vaccine within 2 weeks prior to entry into the study
13. Body temperature ≥38°C.0 (≥100.4° F) and/or acute illness within 3 days of intended study vaccination,
14. Body mass index (BMI) ≥ 35 kg/m2,
15. History of drug or alcohol abuse,
16. Any planned surgery during study period,
17. Individuals conducting the study and their immediate family members,
18. Individuals with behavioral or cognitive impairment or psychiatric diseases.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1393 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (23):
- United States (12):
  - 1 Tatum Highlands Med Ass PLLC, Phoenix, Arizona
  - 5 Broward Research Group Pembroke Pines, Hollywood, Florida
  - 7 Heartland Rsrch Ass LLC, Wichita, Kansas
  - 9 Heartland Research Associates, Wichita, Kansas
  - 2 Mercy Health Research, St Louis, Missouri
  - 3 Saint Louis University, St Louis, Missouri
  - 6 Regional Clinical Research Endwell,, Endwell, New York
  - 4 Benchmark Medical Research, Austin, Texas
  - 12 Tekton Research, Georgetown, Texas
  - 8 J. Lewis Research Inc., Salt Lake City, Utah
  - 10 Foothill Family Clinic, South Cottonwood Heights, Utah
  - 11 Jordan River Family Medicine, South Jordan, Utah
- Australia (5):
  - 42 Hunter Clinical Research, Newcastle, New South Wales
  - 44 Wesley Research Institute Clinical Trials Center, Auchenflower, Queensland
  - 40 CMAX, Adelaide, South Australia
  - 41 Linear Clinical Research, Nedlands, Western Australia
  - 45 Childrens Clin Rsrch Facility, Perth, Western Australia
- New Zealand (2):
  - 50 Southern Clinical Trials, Beckenham, Christchurch
  - 51 Riccarton Clinic, Riccarton, Christchurch
- Thailand (4):
  - 72 Faculty of Medicine, Chulalongkorn University - Queen Saovabha Memorial Institute, Bangkok
  - 71 Phramongkutklao Hospital, Bangkok
  - 73 Siriraj Clinical Research Ctr, Bangkok
  - 74 Chiang Mai Uni Hospital Clinical Trial Center, Bangkok

REFERENCES:
- [Derived] Frey SE, Shakib S, Chanthavanich P, Richmond P, Smith T, Tantawichien T, Kittel C, Jaehnig P, Mojares Z, Verma B, Kanesa-Thasan N, Hohenboken M. Safety and Immunogenicity of MF59-Adjuvanted Cell Culture-Derived A/H5N1 Subunit Influenza Virus Vaccine: Dose-Finding Clinical Trials in Adults and the Elderly. Open Forum Infect Dis. 2019 Mar 1;6(4):ofz107. doi: 10.1093/ofid/ofz107. eCollection 2019 Apr. PMID 30968056

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1393 subjects were enrolled at 12 centers in the US, 5 centers in Australia, 2 centers in New Zealand and 4 centers in Thailand.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- High Dose: Subjects received 2 injections of a high dose of cell culture-derived adjuvanted monovalent inactivated subunit H5N1 vaccine three weeks apart.
- Low Dose: Subjects received 2 injections of a low dose of cell culture-derived adjuvanted monovalent inactivated subunit H5N1 vaccine three weeks apart.
Period: Overall Study
Arm/Group | High Dose | Low Dose
Started | 700 | 693
Completed | 676 | 676
Not Completed | 24 | 17
Not completed — Administrative Reason | 5 | 5
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 1 | 3
Not completed — Unclassified | 2 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 14 | 5

BASELINE CHARACTERISTICS:
Population: Analysis was done on All Enrolled population.
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose | Low Dose | Total
Number analyzed (Participants) | 700 | 693 | 1393
Age, Continuous [Mean (Standard Deviation); unit: year] | 71.2 (5.1) | 70.7 (4.7) | 71.0 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  FEMALE | 407 | 418 | 825
  MALE | 293 | 275 | 568

OUTCOME MEASURES:

1. Primary Outcome: The Percentages Of Subjects Achieving Hemagglutination Inhibition (HI) Titers ≥40 Against A/H5N1 Strain.
Description: The optimal aH5N1c vaccine formulation was evaluated in terms of percentages of subjects achieving HI titers ≥40 against homologous A/H5N1 strain, three weeks after second vaccination with either low dose or high dose of aH5N1c vaccine, according to the Center for Biologics Evaluation and Research (CBER) criterion.
  The CBER criterion for the elderly population is met if the lower limit of the two-sided 95% confidence interval (CI) for the percentages of subjects achieving HI titer ≥40 meets or exceeds 60%.
Time Frame: Baseline (day 1) and Three weeks after 2nd vaccination (day 43)
Population: Analysis was done on the Full Analysis Set (FAS) i.e., subjects who actually receive at least one dose of study vaccination and provide at least one evaluable serum sample both before (baseline) and after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 693 | 683
Percentages of subjects
  Day 1 | 12 [10 to 15] | 10 [8 to 12]
  Day 43 (N=673,664) | 81 [78 to 84] | 63 [59 to 66]

2. Primary Outcome: The Percentages Of Subjects Achieving Seroconversion Against A/H5N1 Strain.
Description: Immunogenicity was measured in terms of the percentages of subjects achieving seroconversion or significant increase in HI titer against the vaccine strain, three weeks after receiving two injections of low dose or high dose of aH5N1c vaccine according to the CBER criterion.
  Seroconversion is defined as, a postvaccination titer ≥40 in subjects with a prevaccination HI titer <10; or in subjects with prevaccination HI titer ≥10, a minimum four-fold rise in postvaccination HI antibody titer.
  The CBER criterion for the elderly population is met if the lower limit of the two-sided 95% CI for the percentages of subjects achieving seroconversion for HI antibody titer meets or exceeds 30%.
Time Frame: Three weeks after 2nd vaccination (day 43)
Population: This analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 673 | 664
Percentages of subjects | 74 [70 to 77] | 52 [48 to 56]

3. Primary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events, After Any Vaccination.
Description: Safety was assessed as the number of subjects who reported solicited local and systemic adverse events following vaccination with either low or high dose of aH5N1c vaccine.
Time Frame: From day 1 through day 7 after any vaccination.
Population: Analysis was done on the solicited safety population, i.e. All subjects in the exposed set with solicited (local/systemic) AE data..
Measure: Number; unit: Number of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 693 | 683
Number of subjects
  Any Local | 314 | 212
  Injection site Erythema (N=693,681) | 17 | 5
  Injection site Induration (N=693,683) | 20 | 11
  Injection site Ecchymosis (N=692,682) | 7 | 10
  Injection site Pain (N=693,681) | 309 | 203
  Any Systemic | 250 | 228
  Nausea (N=692,681) | 45 | 44
  Myalgia (N=691,681) | 91 | 85
  Arthralgia (N=692,681) | 65 | 69
  Headache (N=692,678) | 92 | 89
  Fatigue (N=692,681) | 116 | 112
  Loss of Appetite (N=683,673) | 40 | 42
  Malaise (N=692,680) | 116 | 117
  Fever (≥38°C; N=693,681) | 16 | 4
  Prevention of Pain and (or) Fever (N=691,682) | 18 | 26
  Treatment of Pain and (or) Fever (N=691,682) | 56 | 46

4. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Any Vaccination.
Description: Safety was assessed using the number of subjects who reported any unsolicited adverse events, adverse events possibly or probably related to study vaccine, serious adverse events (SAEs), new onset of chronic diseases (NOCDs), medically attended AEs, AEs of special interest (AESIs), AEs leading to withdrawal from study following vaccination with aH5N1c vaccine
Time Frame: Day 1 through day 387 after any vaccination
Population: Analysis was done unsolicited safety population, i.e. subjects in the exposed set with unsolicited AE data.
Measure: Number; unit: Number of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 694 | 686
Number of subjects
  Any AEs (Day 1 to 22; N=694,685) | 147 | 149
  At least possibly related AEs(Day1to22;N=694,685) | 56 | 61
  Any AEs (Day 23 to 43; N=689,681) | 101 | 123
  At least possibly related AEs(Day23to43;N=689,681) | 21 | 37
  Any SAEs | 43 | 53
  Deaths | 1 | 1
  Medically attended AEs | 383 | 373
  Premature withdrawal from study | 1 | 1
  AESIs | 2 | 0
  NOCD | 108 | 92

5. Secondary Outcome: Geometric Mean Ratios (GMR) Against A/H5N1 Strain Following 2-dose Vaccination Schedule of Either Low Dose or High Dose aH5N1c Vaccine.
Description: Immunogenicity was measured as the GMR. The ratio of postvaccination to prevaccination HI geometric mean titers (GMTs) is reported.
  The criterion is met according to the European Committee for Medicinal Products for Human Use (CHMP) criterion if the geometric mean increase GMR (day 43/day 1) in HI antibody titer is >2.0 for subjects >60 years of age.
Time Frame: Day 1; day 22; day 43 and day 387
Population: Analysis was done on the FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 681 | 673
Ratio
  A/H5N1 (Day22/Day1) | 3.21 [2.85 to 3.62] | 2.01 [1.78 to 2.26]
  A/H5N1 (Day43/Day1; N=673,664) | 16 [14 to 18] | 5.72 [4.94 to 6.63]
  A/H5N1 (Day387/Day1; N=658,651) | 1.97 [1.79 to 2.17] | 1.3 [1.18 to 1.44]

6. Secondary Outcome: Percentages Of Subjects With HI Titers ≥40 Against A/H5N1 Strain
Description: Immunogenicity was assessed in terms of percentage of subjects achieving HI titers >40, three weeks after second vaccination with aH5N1c according to the CHMP criterion.
  The European Licensure (CHMP) criterion is met if the percentage of subjects achieving HI titers ≥40 is >60%.
Time Frame: Day 1, day 22, day 43 and day 387.
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 693 | 683
Percentages of subjects
  Day 1 | 12 [10 to 15] | 10 [8 to 12]
  Day 22 (N=681,673) | 49 [45 to 52] | 32 [28 to 35]
  Day 43 (N=673,664) | 81 [78 to 84] | 63 [59 to 66]
  Day 387 (N=658,651) | 35 [31 to 39] | 16 [13 to 19]

7. Secondary Outcome: The Percentages Of Subjects Achieving Seroconversion Against A/H5N1 Strain
Description: Immunogenicity was assessed in terms of percentages of subjects achieving seroconversion in HI titers, three weeks after receiving two injections of either low dose or high dose aH5N1c vaccine according to the CHMP criterion.
  Seroconversion is defined as a postvaccination titer ≥40 in subjects with a prevaccination HI titer <10; or in subjects with prevaccination HI titer ≥10, a minimum four-fold rise in postvaccination HI antibody titer.
  The criterion is met according to the European (CHMP) guideline if the percentage of subjects achieving seroconversion is >30%.
Time Frame: Day 22, day 43 and day 387
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 681 | 673
Percentages of subjects
  Day 22 | 36 [32 to 40] | 21 [18 to 25]
  Day 43 (N=673,664) | 74 [70 to 77] | 52 [48 to 56]
  Day 387 (N=658,651) | 23 [20 to 27] | 10 [8 to 12]

ADVERSE EVENTS:
Time Frame: Solicited local and systemic adverse events were collected from day 1 to 7. Unsolicited AEs (other than SAEs) and SAEs were collected from day 1 to 387.
Description: All Solicited AEs-systematic assessment and all unsolicited AEs-non-systematic assessment.
  Type II reactions are reported for solicited AEs. Total number of subjects enrolled was - High dose: 700 and Low dose: 693. Total number of subjects who received a study vaccination and included in safety set was - High dose: 699 and Low dose: 689
Groups:
- High Dose: Subjects received 2 injections of a high dose MF59 adjuvanted cell-culture derived monovalent H5N1 vaccine three weeks apart.
- Low Dose: Subjects received 2 injections of a low dose MF59 adjuvanted cell-culture derived monovalent H5N1 three weeks apart.
- Total: Total of subjects in both high and low dose groups.
Arm/Group | High Dose | Low Dose | Total
Serious Adverse Events (participants affected / at risk) | 43/699 | 51/689 | 94/1388
Other Adverse Events (participants affected / at risk) | 481/699 | 427/689 | 908/1388
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose (N=699) | Low Dose (N=689) | Total (N=1388)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 1 | 2
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 3 | 2 | 5
ATRIAL FLUTTER (Cardiac disorders) | 0 | 2 | 2
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 | 1 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 2 | 3
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 1 | 2
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 1 | 1
PERICARDITIS (Cardiac disorders) | 0 | 1 | 1
SICK SINUS SYNDROME (Cardiac disorders) | 0 | 1 | 1
STRESS CARDIOMYOPATHY (Cardiac disorders) | 1 | 0 | 1
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 | 1 | 1
CATARACT (Eye disorders) | 1 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 1
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 1
DUODENAL ULCER PERFORATION (Gastrointestinal disorders) | 0 | 1 | 1
ENTERITIS (Gastrointestinal disorders) | 0 | 1 | 1
EPIPLOIC APPENDAGITIS (Gastrointestinal disorders) | 0 | 1 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 2 | 2
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 1
CHEST DISCOMFORT (General disorders) | 0 | 1 | 1
CHEST PAIN (General disorders) | 1 | 2 | 3
PYREXIA (General disorders) | 0 | 2 | 2
CHOLECYSTITIS (Hepatobiliary disorders) | 3 | 0 | 3
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 | 0 | 1
ANAL ABSCESS (Infections and infestations) | 0 | 1 | 1
DIVERTICULITIS (Infections and infestations) | 0 | 1 | 1
MENINGITIS VIRAL (Infections and infestations) | 1 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 1 | 1
POST PROCEDURAL INFECTION (Infections and infestations) | 0 | 1 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 2 | 2
WOUND INFECTION (Infections and infestations) | 1 | 0 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 2 | 2
CONCUSSION (Injury, poisoning and procedural complications) | 1 | 0 | 1
FALL (Injury, poisoning and procedural complications) | 0 | 1 | 1
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 | 0 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 2 | 2
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 1
TRAUMATIC HAEMOTHORAX (Injury, poisoning and procedural complications) | 0 | 1 | 1
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
BONE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
ENDOMETRIAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
LENTIGO MALIGNA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
MALIGNANT MELANOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 4
BASAL GANGLIA INFARCTION (Nervous system disorders) | 1 | 0 | 1
BRAIN STEM INFARCTION (Nervous system disorders) | 1 | 0 | 1
CAROTID ARTERY DISEASE (Nervous system disorders) | 0 | 1 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 1 | 1 | 2
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 1 | 2
EMBOLIC STROKE (Nervous system disorders) | 1 | 0 | 1
HEADACHE (Nervous system disorders) | 0 | 1 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 0 | 1
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 1 | 1
SYNCOPE (Nervous system disorders) | 0 | 3 | 3
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 2 | 2
VIITH NERVE PARALYSIS (Nervous system disorders) | 1 | 0 | 1
GRIEF REACTION (Psychiatric disorders) | 1 | 0 | 1
SUICIDAL IDEATION (Psychiatric disorders) | 1 | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 0 | 1
RENAL COLIC (Renal and urinary disorders) | 0 | 1 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0 | 1
RECTOCELE (Reproductive system and breast disorders) | 0 | 1 | 1
UTERINE POLYP (Reproductive system and breast disorders) | 0 | 1 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 | 0 | 1
AORTIC ANEURYSM (Vascular disorders) | 1 | 0 | 1
AORTIC STENOSIS (Vascular disorders) | 0 | 1 | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose (N=699) | Low Dose (N=689) | Total (N=1388)
NAUSEA (Gastrointestinal disorders) | 48 | 47 | 95
FATIGUE (General disorders) | 119 | 117 | 236
INJECTION SITE PAIN (General disorders) | 317 | 210 | 527
MALAISE (General disorders) | 116 | 119 | 235
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 32 | 36 | 68
EATING DISORDER (Psychiatric disorders) | 40 | 43 | 83
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 87 | 87 | 174
MYALGIA (Musculoskeletal and connective tissue disorders) | 103 | 93 | 196
HEADACHE (Nervous system disorders) | 108 | 104 | 212

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No